CLINICAL TRIAL: NCT07122934
Title: Posterior Circulation Clot Burden Score (Pc-CBS) Predicts Clinical Outcome After Acute Ischemic Stroke Related to Posterior Circulation Occlusions : An Externally Validated Radiological Score
Acronym: PC-CBS
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Collaborators: Insel Gruppe AG, University Hospital Bern (Other); Hospital de Egas Moniz (Other); University Hospital Heidelberg (Other); IRCCS Istituto delle Scienze Neurologiche di Bologna (Other); The University of Texas Health Science Center, Houston (Other); Azienda Ospedaliero-Universitaria di Modena (Other); Hospital Vall d'Hebron (Other); Boston University (Other); Università degli Studi di Brescia (Other); Medical University of Graz (Other); Hôpital Rothschild (Other); Medical University of Vienna (Other); Hebrew University of Jerusalem (Other); Michigan State University (Other); Medical University Innsbruck (Other); Ludwig-Maximilians - University of Munich (Other); Ospedale Policlinico San Martino (Other); EOC Lugano CH (Unknown); University Hospital, Basel, Switzerland (Other); Aristotle University Of Thessaloniki (Other); Technische Universität Dresden (Other)
Responsible Party: Principal Investigator, Dr. med. Alexander Salerno, MD-PhD, Senior registrar, Centre Hospitalier Universitaire Vaudois
Other Study IDs: PC-CBS
Record Dates: First submitted 2025-08-08; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Acute Ischemic Stroke; Posterior Circulation Brain Infarction; Arterial Occlusion Disease
MeSH Terms: conditions — Ischemic Stroke; Brain Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Development and Internal validation cohort
  Interventions: Diagnostic Test: Assessment of cervico-cerebral arterial occlusion pattern
- External validation cohort
  Interventions: Diagnostic Test: Assessment of cervico-cerebral arterial occlusion pattern

INTERVENTIONS:
Diagnostic Test: Assessment of cervico-cerebral arterial occlusion pattern — Assessment of cervico-cerebral arterial occlusion pattern for the development of a radiological score

SUMMARY:
Posterior circulation strokes (PCS) represent ~30% of all ischemic strokes, but existing prognostic tools are limited, especially for non-basilar artery occlusions. Accurate early outcome prediction may aid treatment decisions and clinical trial design. We developed and externally validated the Posterior Circulation Clot Burden Score (PC-CBS), a radiological tool to predict 3-month functional outcome in acute ischemic stroke due to posterior circulation occlusion.

ELIGIBILITY:
Inclusion Criteria:

* age >18 years old
* admitted within 24h from last known well
* symptomatic arterial occlusion. The following arterial occlusions were eligible for inclusion: the extracranial vertebral artery between the V0 and V3 segments; the intracranial portion of the vertebral artery; the basilar artery either in its proximal, mid and/or distal segment, the P1 and/or the P2 segments of the posterior cerebral artery.

Exclusion Criteria:

* simultaneous clinical and/or radiological strokes in the posterior and anterior circulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from an acute ischemic stroke (AIS) clinically and/or radiologically attributable to a posterior circulation arterial occlusion
Sampling Method: Non-Probability Sample
Enrollment: 1828 (Actual)
Dates: Start 2003-02-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2025-08-08 (Actual)

PRIMARY OUTCOMES:
Modified rankin scale at three months | 3 months